CLINICAL TRIAL: NCT01753531
Title: A Multicenter Performance Evaluation for the Ultra Influenza A&B Test Using Nasal Swabs
Brief Title: Clinical Performance Study of the Ultra Influenza A&B Test Using Nasal Swabs for Identifying Subjects Who Are Infected With the Influenza Virus Strain Type A or Type B
Status: Completed | Type: Observational
Sponsor: Sekisui Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CAP-199
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Influenza, Human
Keywords: Ultra Influenza A and B; Influenza Type A; Influenza Type B; Flu; Sekisui Diagnostics
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swab specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Flu Symptoms
  Interventions: Device: Flu Symptoms

INTERVENTIONS:
Device: Flu Symptoms

SUMMARY:
The clinical performance of the Ultra Influenza A&B Test will be demonstrated during a clinical trial in which prospectively collected nasal swabs are used in identifying subjects who are infected with the influenza virus strain type A or type B. The Ultra Influenza A&B Test qualitative results will be compared to "Gold Standard" viral culture with Direct Fluorescent Antibody (DFA) confirmation techniques using nasal swabs collected from symptomatic subjects. The Ultra Influenza A&B Test will be performed at Clinical Laboratory Improvement Amendments (CLIA) waived sites by untrained intended users (e.g. nurses, physician assistants, medical assistants, etc.). For viral culture testing with DFA confirmation testing, nasal swab specimen testing will be performed by a designated reference laboratory.

ELIGIBILITY:
Inclusion Criteria:

* The subject may be of any age and either gender.
* Preliminary assessment of the subject by the Investigator/designee should be suggestive of influenza virus infection. Subject should present with an influenza-like febrile respiratory illness defined as (1) presentation within the last 48 hours of developing a subjective feeling of being feverish and/or a temperature recorded at the clinic within the last 48 hours of greater than or equal to 100.5 F and (2) at least two of the following symptoms: cough, nasal congestion, rhinorrhea, sore throat, headache, myalgia.
* Written informed consent must be obtained prior to study enrollment.

  1. A subject who is 18 years or older must be willing to give written informed consent and must agree to comply with study procedures.
  2. The legal authorized representative of a subject who is under the age of 18 must give written informed consent and agree to comply with study procedures. Active written assent should be obtained from children of appropriate intellectual age (as defined by the IRB).

Exclusion Criteria:

* The subject underwent a nasal wash/aspirate as part of standard-of-care testing during this study visit.
* The subject is undergoing treatment currently and/or within the past 7 days of the study visit with a nasally administered influenza vaccine (FluMist) or with anti-viral medication, which may include but is not limited to Amantadine (Symmetrel), Rimantadine (Flumadine), Zanamivir (Relenza), Oseltamivir (Tamiflu) or Ribavirin.
* The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug or device, including either treatment or therapy.
* The subject has previously participated in this research study.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects presenting with symptoms suggestive of influenza virus infection will be enrolled from geographically diverse CLIA Waived Intended Users (Physicians office laboratories, clinics or equivalents)
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Identify subjects who are infected with the virus strain type A or type B | 6 months
  Characterize the performance of the Ultra Influenza A&B Test and to identify subjects who are infected with the influenza virus strain type A or type B. Performance data generated will support a 510k submission to FDA for clearance of the assay.

SECONDARY OUTCOMES:
Demonstrate the ability of untrained intended users to effectively run and read the Ultra Influenza A&B Test with insignificant risk of erroneous results. | 6 months
  Demonstrate the ability of untrained intended users to effectively run and read the Ultra Influenza A&B Test with insignificant risk of erroneous results. Qualitative results obtained using the Ultra Influenza A&B Test will be compared to viral culture with direct fluorescent antibody (DFA) confirmation testing on specimens collected during this study. Data demonstrating ease of use will support a request to FDA for CLIA waived categorization of the assay.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Rosen, MD, Principal Investigator — Ardmore Family Practice
Locations (3):
- United States (3):
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - Hill Country Medical Associates, New Braunfels, Texas